CLINICAL TRIAL: NCT03768505
Title: A Multicenter, Open Label Single-Arm, Phase 2 Study of Zandelisib (ME-401) in Subjects With Follicular Lymphoma and Marginal Zone Lymphoma After Failure of Two or More Prior Systemic Therapies (The TIDAL Study)
Brief Title: Zandelisib (ME-401) in Subjects With Follicular Lymphoma or Marginal Zone Lymphoma After Failure of Two or More Prior Therapies (TIDAL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: discontinuation of zandelisib program
Sponsor: MEI Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-401-003; 2018-002896-17 (EudraCT Number)
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2022-12

CONDITIONS: Follicular Lymphoma (FL); Non Hodgkin Lymphoma; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone | interventions — ME-401

STUDY DESIGN:
Intervention Model Description: Treatment with Zandelisib (ME-401) (60 mg) given orally once a day on an intermittent schedule
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zandelisib (ME-401) open label (Experimental): Subjects with relapsed/refractory FL or MZL will be administered 60 mg of ME-401 orally, once a day on an intermittent schedule (IS).
  Interventions: Drug: Zandelisib (ME-401)

INTERVENTIONS:
Drug: Zandelisib (ME-401) — Zandelisib (ME-401) 60 mg

SUMMARY:
This is the study of the PI3Kδ inhibitor Zandelisib (ME-401) in subjects with relapsed/refractory follicular lymphoma or marginal zone lymphoma after failure of at least 2 prior lines of systemic therapy

DETAILED DESCRIPTION:
This is a global, multicenter open-label, single-arm, Phase 2 study of the PI3Kδ inhibitor Zandelisib (ME-401) in subjects with relapsed/refractory follicular lymphoma or marginal zone lymphoma after failure of at least 2 prior lines of systemic therapy which must have included an anti-CD20 antibody and chemotherapy with an alkylating agent or a purine analogue.

Approximately 180 subjects will be enrolled and treated with Zandelisib (ME-401) on the intermittent schedule.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis as defined in the World Health Organization (WHO) classification scheme

  1. Follicular Lymphoma (FL) limited to Grade 1,2 or 3a or
  2. Marginal Zone Lymphoma (MZL) including nodal, extranodal and splenic MZL
* Subjects that have had progression of disease or had no response to therapy after at least 2 prior systemic therapies for FL or MZL
* Age ≥ 18
* At least one bi-dimensionally measurable nodal lesion > 1.5 cm in its longest diameter by computed tomography (CT) scan as defined by the Lugano Classification
* Adequate hematologic, renal and hepatic parameters at screening unless abnormal values are due to FL per Investigator assessment
* QT-interval corrected according to Fridericia's formula (QTcF) ≤ 450 milliseconds (msec);
* Left ventricular ejection fraction (LVEF) ≥ 45%

Exclusion Criteria:

* Histologically confirmed FL Grade 3b transformation from FL to an aggressive lymphoma
* Known lymphomatous involvement of the central nervous system
* Uncontrolled clinically significant illness
* Ongoing or history of drug-induced pneumonitis
* History of clinically significant cardiovascular abnormalities
* History of clinically significant GI conditions
* Known history of, or active HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (115):
- United States (34):
  - Oncology Institute of Hope and Innovation, Tucson, Arizona
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Tower Hematology Oncology, Beverly Hills, California
  - The Oncology Institute of Hope and Innovation, Downey, California
  - Sharp Memorial Hospital, San Diego, California
  - H. Lee Moffit Cancer Center, Tampa, Florida
  - Cleveland Clinic-Florida, Weston, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Health & Hospitals Corporation, Niles, Illinois
  - Investigative Clinical Research of Indiana LLC, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Medical School, Ann Arbor, Michigan
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - The Oncology Institute of Hope and Innovation, Henderson, Nevada
  - Memorial Sloan Kettering, Basking Ridge, New Jersey
  - Memorial Sloan Kettering, Middletown, New Jersey
  - Memorial Sloan Kettering, Montvale, New Jersey
  - San Juan Oncology, Farmington, New Mexico
  - Memorial Sloan Kettering, Commack, New York
  - Memorial Sloan Kettering, Harrison, New York
  - Clinical Research Alliance, Lake Success, New York
  - Memorial Sloan Kettering, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Memorial Sloan Kettering, Uniondale, New York
  - Duke Cancer Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - Renovatio Clinical, Houston, Texas
  - Swedish Cancer Institute, Edmonds, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Medical Oncology Associates PS, Spokane, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
- Australia (3):
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - The Perth Blood Institute, West Perth, Western Australia
  - Liverpool Hospital, Sydney
- Austria (2):
  - Kepler Universitatsklinikum GmBH, Linz
  - Medical University of Vienna, Vienna
- Belgium (4):
  - AZ Sint-Jan Brugge-Oostende, Bruges
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
- France (6):
  - C H de la Cote Basque, Service d'Hematologie, Bayonne
  - CHD Vendee, Onco-hematologie, La Roche-sur-Yon
  - Centre Hospitalier du Mans, Le Mans
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre Hospitalier Universitaire (CHU) de Poitiers - Hôpital de la Miletrie, Poitiers
  - Institut Gustave Roussy, Villejuif
- Germany (6):
  - Klinikum Mutterhaus Feldstr, Trier, Rhineland-Palatinate
  - Hamatologisch-Onkolgische Praxis, Nordheim, Stolberg
  - Universitatsklinikum Halle, Halle
  - Munich Municipal Hospital, Munich
  - Universitatsklinikum Munster, Münster
  - Universitatsklinikum Ulm, Ulm
- Italy (11):
  - Centro di Riferimento Oncologico di Aviano (CRO) IRCCS, Aviano
  - Policlinico Sant'Orsola Malpighi, Bologna
  - IRCCS AOU Policlinico San Martino, Genova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori I.R.S.T., Meldola
  - UOC Oncoematologia, Napoli
  - Ospedale Santa Maria delle Croci, Ravenna
  - Infermi Hospital Rimini, Rimini
  - Universita Cattolica del Sacro Cuore, Roma
  - IRCCS Regina Elena National Cancer Institute, Rome
  - Azienda Ospedaliera Santa Maria, Terni
  - Ospedale DellAngelo Di Mestre Umberto I, Venice
- New Zealand (2):
  - North Shore Hospital, Auckland
  - Southern District Hospital, Dunedin
- Poland (6):
  - Szpital Uniwersytecki nr 2 im., Bydgoszcz
  - Pratia MCM Krakow, Krakow
  - ojewodzkie Wielospecjalistyczne Centrum, Lodz
  - Primary Specialty Oncology, Warsaw
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Dolnoslaskie Centrum Transplantacji Komorkowych z Krajowym Bankiem Dawcow Szpiku, Wroclaw
- South Korea (9):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - The Catholic University of Korea-Seoul St. Marys Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (13):
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari Mutua Terrasa, Barcelona
  - ICO-Hospital Duran i Reynals, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Quiron Salud Madrid, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Clinico de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Virgen del Rocio, Seville
  - Miguel Servet Hospital, Zaragoza
- Ente Ospedaliero Cantonale (EOC), Bellinzona, Switzerland
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi-Mei Medical Center, Liouying, Tainan
  - National Taiwan University Hospital NTUH, Taipei
- United Kingdom (14):
  - North Wales Cancer Treatment Centre, Glan Clwyd Hospital, Rhyl, Denbighire
  - Royal Marsden Hospital, London, Sutton
  - Nottingham University Hospital, Nottingham, UK
  - Belfast Health and Social Care Trust - Belfast City Hospital, Belfast
  - Royal Cornwall Hospital, Cornwell
  - e Clatterbridge Cancer Centre, Liverpool
  - Royal Liverpool University Hospital, Liverpool
  - Lewisham and Greenwich University Hospital Lewisham, London
  - St George's Hospital, London
  - Centre for Haematology, Imperial College London, London
  - The Christie NHS Foundation Trust, Manchester
  - Norfolk and Norwich University Hospital NHS Foundation Trust, Norwich
  - Oxford University Hospitals, Oxford
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2 study was open from June 2019 to March 2023 at 124 investigational sites in the United States, United Kingdom, Spain, New Zealand, Austria, South Korea, Belgium, Taiwan, Poland, Italy, Australia, France, Germany. This study was closed prematurely for business reasons . A total of 169 subjects were enrolled. The reasons for subjects not completing the study are listed below. The majority was due to study closure by sponsor.
Groups:
- Zandelisib (ME-401) Open Label: Subjects with relapsed/refractory FL or MZL were administered 60 mg of ME-401 orally, once a day on an intermittent schedule (IS).
  Zandelisib (ME-401): Zandelisib (ME-401) 60 mg
Period: Overall Study
Arm/Group | Zandelisib (ME-401) Open Label
Started | 169
Completed | 0
Not Completed | 169
Not completed — sponsor decision | 76
Not completed — Death | 35
Not completed — Other -Various | 30
Not completed — Withdrawal by Subject | 22
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Zandelisib (ME-401) Open Label
Number analyzed (Participants) | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 79
  >=65 years | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 144
  Unknown or Not Reported | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 129
  More than one race | 0
  Unknown or Not Reported | 15
Region of Enrollment [Number; unit: participants]
  United States | 26
  United Kingdom | 34
  Spain | 8
  New Zealand | 5
  Austria | 3
  South Korea | 15
  Belgium | 8
  Taiwan | 7
  Poland | 18
  Italy | 21
  Australia | 8
  France | 12
  Germany | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of ME-401 in Relapsed or Refractory FL or MZL
Description: ORR is measured as the proportion of subjects achieving the best response rating of CR or PR prior to first PD
Time Frame: 3 years 9 months
Population: A company decision was made to terminate all Zandelisib studies early due to business reasons including this Phase 2 study. Due to the study being terminated early, no data was collected to analyze ORR
Arm/Group | Zandelisib (ME-401) Open Label
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response will be measured as the time from documentation from CR or PR to time of disease progression
Time Frame: 3 years 9 months
Population: A company decision was made to terminate all Zandelisib studies early due to business reasons including this Phase 2 study. Due to the study being terminated early, no data was collected to analyze DOR
Arm/Group | Zandelisib (ME-401) Open Label
Number analyzed (Participants) | 0

3. Secondary Outcome: Complete Response (CR) Rate
Description: Complete response rate will be measured by the number of subjects that achieve CR
Time Frame: 3 years 9 months
Population: A company decision was made to terminate all Zandelisib studies early due to business reasons including this Phase 2 study. Due to the study being terminated early, no data was collected to analyze CR
Arm/Group | Zandelisib (ME-401) Open Label
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival will be measurement of time from initiation of treatment (Day 1) until disease progression or death
Time Frame: 3 years 9 months
Population: A company decision was made to terminate all Zandelisib studies early due to business reasons including this Phase 2 study. Due to the study being terminated early, no data was collected to analyze PFS.
Arm/Group | Zandelisib (ME-401) Open Label
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival will be measured as the time from initiation of treatment (Day 1) until death
Time Frame: 2 years
Population: Study was terminated early, therefore data was not available to measure OS at time of termination
Arm/Group | Zandelisib (ME-401) Open Label
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Incidence of Treatment Emergent Adverse Events (TEAEs)
Description: The incidence of TEAEs is measured by the proportion of subjects with at least one TEAE.
Time Frame: 3 years 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Zandelisib (ME-401) Open Label
Number analyzed (Participants) | 162
Participants | 162

7. Secondary Outcome: PK of ME-401
Description: The PK of ME-401 will be determined by the peak plasma concentration (Cmax)
Time Frame: 3 years 9 months
Population: A company decision was made to terminate all Zandelisib studies early due to business reasons including this Phase 2 study. Due to the study being terminated early, no data was collected to analyze PK
Arm/Group | Zandelisib (ME-401) Open Label
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs were collected for 3 years 9 months
Arm/Group | Zandelisib (ME-401) Open Label
All-Cause Mortality (participants affected / at risk) | 35/169
Serious Adverse Events (participants affected / at risk) | 69/169
Other Adverse Events (participants affected / at risk) | 162/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zandelisib (ME-401) Open Label (N=169)
Pneumonia (Infections and infestations) | 8 (8)
COVID-19 pneumonia (Infections and infestations) | 6 (6)
COVID-19 (Infections and infestations) | 4 (4)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1)
Aspergillus infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Autoimmune enteropathy (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Mucosal inflammation (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (3)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Uveitis (Eye disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zandelisib (ME-401) Open Label (N=169)
Diarrhoea (Gastrointestinal disorders) | 66 (66)
Nausea (Gastrointestinal disorders) | 38 (38)
Abdominal pain (Gastrointestinal disorders) | 24 (24)
Constipation (Gastrointestinal disorders) | 22 (22)
Vomiting (Gastrointestinal disorders) | 11 (11)
Dyspepsia (Gastrointestinal disorders) | 10 (10)
Stomatitis (Gastrointestinal disorders) | 9 (9)
Colitis (Gastrointestinal disorders) | 6 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Flatulence (Gastrointestinal disorders) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 2 (2)
Eructation (Gastrointestinal disorders) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Melaena (Gastrointestinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 2 (2)
Abdominal rigidity (Gastrointestinal disorders) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 1 (1)
Autoimmune enteropathy (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 (1)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 23 (23)
Urinary tract infection (Infections and infestations) | 10 (10)
Pneumonia (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 10 (10)
Herpes zoster (Infections and infestations) | 9 (9)
Cytomegalovirus infection (Infections and infestations) | 7 (7)
Asymptomatic COVID-19 (Infections and infestations) | 6 (6)
Bronchitis (Infections and infestations) | 6 (6)
COVID-19 pneumonia (Infections and infestations) | 2 (2)
Cytomegalovirus infection reactivation (Infections and infestations) | 5 (5)
Herpes simplex (Infections and infestations) | 5 (5)
Sinusitis (Infections and infestations) | 5 (5)
Nasopharyngitis (Infections and infestations) | 4 (4)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 (3)
Candida infection (Infections and infestations) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 3 (3)
Diverticulitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1)
Bacterial diarrhoea (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Cytomegalovirus gastroenteritis (Infections and infestations) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Oral viral infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 30 (30)
Pyrexia (General disorders) | 26 (26)
Asthenia (General disorders) | 14 (14)
Oedema peripheral (General disorders) | 10 (10)
Chest pain (General disorders) | 4 (4)
Mucosal inflammation (General disorders) | 4 (4)
Chills (General disorders) | 3 (3)
Influenza like illness (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (3)
Chest discomfort (General disorders) | 2 (2)
Gait disturbance (General disorders) | 2 (2)
Inflammation (General disorders) | 2 (2)
Cyst (General disorders) | 1 (1)
Discomfort (General disorders) | 1 (1)
Drug intolerance (General disorders) | 1 (1)
Hyperthermia (General disorders) | 1 (1)
Injection site rash (General disorders) | 1 (1)
Localised oedema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Swelling face (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 21 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (13)
Night sweats (Skin and subcutaneous tissue disorders) | 5 (5)
Rash erythematous (Skin and subcutaneous tissue disorders) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Granuloma annulare (Skin and subcutaneous tissue disorders) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1)
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 19 (19)
Weight decreased (Investigations) | 16 (16)
ALT increased (Investigations) | 14 (14)
AST increased (Investigations) | 13 (13)
Blood creatinine increased (Investigations) | 11 (11)
Platelet count decreased (Investigations) | 8 (8)
Blood lactate dehydrogenase increased (Investigations) | 8 (8)
White blood cell count decreased (Investigations) | 8 (8)
Lymphocyte count decreased (Investigations) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 4 (4)
C-reactive protein increased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 3 (3)
Blood cholesterol increased (Investigations) | 2 (2)
Blood lactate dehydrogenase (Investigations) | 2 (2)
Cytomegalovirus test positive (Investigations) | 2 (2)
Lymphocyte count increased (Investigations) | 2 (2)
AST/ALT ratio abnormal (Investigations) | 1 (1)
Aspartate aminotransferase (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood creatinine decreased (Investigations) | 1 (1)
Blood immunoglobulin G decreased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Prothrombin time shortened (Investigations) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Vitamin D decreased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 28 (28)
Anaemia (Blood and lymphatic system disorders) | 20 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (16)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 23 (23)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4)
Appetite disorder (Metabolism and nutrition disorders) | 2 (2)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Overweight (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (24)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 18 (18)
Dizziness (Nervous system disorders) | 12 (12)
Paraesthesia (Nervous system disorders) | 5 (5)
Memory impairment (Nervous system disorders) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 3 (3)
Lethargy (Nervous system disorders) | 3 (3)
Balance disorder (Nervous system disorders) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2)
Taste disorder (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Monoparesis (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 5 (5)
Haematuria (Renal and urinary disorders) | 5 (5)
Pollakiuria (Renal and urinary disorders) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal impairment (Renal and urinary disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Glycosuria (Renal and urinary disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Palpitations (Cardiac disorders) | 3 (3)
Ventricular extrasystoles (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Hyperdynamic left ventricle (Cardiac disorders) | 1 (1)
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (9)
Depression (Psychiatric disorders) | 5 (5)
Anxiety (Psychiatric disorders) | 4 (4)
Affect lability (Psychiatric disorders) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypertension (Vascular disorders) | 7 (7)
Hypotension (Vascular disorders) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Raynaud's phenomenon (Vascular disorders) | 2 (2)
Hot flush (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Hepatotoxicity (Hepatobiliary disorders) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 1 (1)
Otolithiasis (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Ocular discomfort (Eye disorders) | 2 (2)
Blepharitis (Eye disorders) | 1 (1)
Eye discharge (Eye disorders) | 1 (1)
Eye haematoma (Eye disorders) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1)
Punctate keratitis (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1)
Pelvic discomfort (Reproductive system and breast disorders) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Ichthyosis (Congenital, familial and genetic disorders) | 1 (1)
Device failure (Product Issues) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed prematurely for business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This study was terminated early however, each PI has a CDA in place that restricts them from discussing any results of the clinical study at a scientific meeting or any other public or private forum or to publish in a scientific or academic journal the results of the clinical study without the approval of the Sponsor Company (MEI Pharma Inc.).

DOCUMENTS (2):
  • Study Protocol (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03768505/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT03768505/SAP_001.pdf